CLINICAL TRIAL: NCT01457235
Title: The Effects of Cognitive Remediation on Cognitive Function in Remitted Bipolar Disorder - a Proof of Concept Study (REMEDI)
Brief Title: The Effects of Cognitive Remediation on Cognitive Function in Remitted Bipolar Disorder - a Proof of Concept Study
Acronym: REMEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Kamilla Miskowiak, Psychologist, Dr., Psychiatric Centre Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-1-2010-039
Record Dates: First submitted 2011-10-10; First posted 2011-10-21 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Cognitive Remediation; Cognition; Cognitive function; Mood disorders; Affective disorders
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Group (Active Comparator): This group receives cognitive remediation in groups (each group consisting of 6-8 subjects)
  Interventions: Other: Cognitive Remediation
- Waiting List (No Intervention): Patients randomized to the waiting list group continues standard treatment and will be offered a course of cognitive remediation upon completion of participation provided that they still meet the inclusion criteria.

INTERVENTIONS:
Other: Cognitive Remediation — All subjects will complete an MR brain scan, blood test, saliva test, and a neuropsychological battery of manual and computerised tests at baseline, at week 12 (end of active treatment) and week 26 (follow-up). Subjects randomly allocated to an active group will participate in a 12-week group-based cognitive remediation programme once a week for two hours. The waiting list group continues treatment as usual.
  Arms: Active Group

SUMMARY:
Cognitive remediation (CR) is a new psychological treatment, which aims to improve cognitive function and coping skills. Several studies have recently demonstrated that CR improves cognitive and occupational function in patients with schizophrenia and with depression (e.g. Wykes et al 2007, Elgamal et al 2007). However, it is unclear whether CR improves cognitive and socio-occupational function in individuals with bipolar disorder (BD) and, if so, what impact this might have on these people's abilities in terms of work, coping strategies, quality of life, and everyday safety.

The aim of the present PhD study is to investigate if CR has beneficial effects on cognitive and socio-occupational function in patients with previous mania and depression who experience persistent cognitive difficulties. Such effects would suggest implementation of CR in future treatment of bipolar disorder in order to facilitate the patients' ability to cope with the responsibilities related to work and everyday life. The hypotheses of the present study are that CR (in comparison to standard treatment) will 1) improve verbal learning and recall; and 2) improve sustained attention, executive function and psychosocial function.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder in complete or partial remission (Hamilton Depression Rating Scale score of max 14 and Young Mania Scale score of max 14)
* Subjective complaints of moderate to severe cognitive problems on the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) (Fava et al 2006) (score at least 4 on at least 2 domains)

Exclusion Criteria:

* Current ECT treatment
* Drug and/or alcohol abuse
* Schizophrenia
* Significant risk of suicide
* Use of benzodiazepines equivalent to more than 22,5 milligrams of Alopam

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Enhance verbal learning and memory as reflected by increase in Rey Auditory Verbal Learning Test (RAVLT) total learning scores and recall | Baseline and weeks 12 and 26
  We expect a clinically relevant difference in the change between groups to be at least 4 points on RAVLT total scores.

SECONDARY OUTCOMES:
Improve sustained attention | Baseline and weeks 12 and 26
  Increase total scores of sustained attention measured with the Rapid Visual Information Processing (RVP) test from baseline to post treatment (week 12)
Improve executive function | Baseline and weeks 12 and 26
  Increase total scores of executive function measured with the Trail Making Test (TMT) part B from baseline to post treatment (week 12)
Increase psychosocial function | Baseline and weeks 12 and 26
  Increase psychosocial function measured with Functional Assessment Short Test (FAST) total scores from baseline to post treatment (week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla W Miskowiak, Dr, Principal Investigator — Psychiatric Centre Copenhagen, Rigshospitalet, Denmark
Locations (1):
- Psychiatric Centre Copenhagen, Rigshospitalet, Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Demant KM, Vinberg M, Kessing LV, Miskowiak KW. Effects of Short-Term Cognitive Remediation on Cognitive Dysfunction in Partially or Fully Remitted Individuals with Bipolar Disorder: Results of a Randomised Controlled Trial. PLoS One. 2015 Jun 12;10(6):e0127955. doi: 10.1371/journal.pone.0127955. eCollection 2015. PMID 26070195
- [Derived] Demant KM, Almer GM, Vinberg M, Kessing LV, Miskowiak KW. Effects of cognitive remediation on cognitive dysfunction in partially or fully remitted patients with bipolar disorder: study protocol for a randomized controlled trial. Trials. 2013 Nov 10;14:378. doi: 10.1186/1745-6215-14-378. PMID 24206639